CLINICAL TRIAL: NCT05011682
Title: The Effect of Nutrition and Medical Therapy on Post-bariatric Hypoglycemia Patients 2-4 Years After a Roux-en-Y Gastric Bypass: a Pilot Study
Brief Title: The Effect of 'Medical Nutrition Therapy' on Post-bariatric Hypoglycemia 2-4 Years After Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/230363
Record Dates: First submitted 2021-08-17; First posted 2021-08-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hypoglycemia; Obesity, Morbid
Keywords: Gastric bypass; Diet therapy; Blood sugar variation; Quality of Life
MeSH Terms: conditions — Hypoglycemia; Obesity, Morbid | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Participants are their own controls. All participants will follow their usual diet in the first 2 weeks, and then during the next 2 weeks the 10-point nutrition plan according to Joslin Diabetes Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Joslin Diabetes Senter nutrition (Experimental): all participants will first follow their own usual diet (2 weeks) and then the Joslin Diabetes Senter nutrition plan (2 weeks)
  Interventions: Behavioral: Regular diet; Behavioral: 10-point nutrition plan

INTERVENTIONS:
Behavioral: Regular diet — participant's usual diet during 2 weeks
Behavioral: 10-point nutrition plan — controlled portions of low glycemic index carbohydrates, avoidance of rapidly absorbed carbohydrates, adjustment of timing of meals and snacks, and attention to personal and cultural barriers to implementation
  Other Names: Joslin Diabetes Senter nutrition plan

SUMMARY:
This is a pilot study to explore the effect of 'medical nutritional therapy' in patients diagnosed with post-bariatric hypoglycemia (PBH), 2-4 years after gastric bypass surgery. The study is largely inspired by the findings presented in the meta-analyses from Joslin Diabetes Center, where a treatment strategy is proposed to reduce the symptoms of PBH. This treatment strategy is mainly based on clinical observations and experience, while there is little or no objective data to support that this strategy improves PBH. The data from this pilot study can then be used to set up larger studies where a conclusion on treatment of PBH may be drawn.

ELIGIBILITY:
Inclusion Criteria:

* patient in Nord-Trøndelag 2-4 years after Roux-en-y gastric bypass surgery
* visits Namsos outpatient clinic for follow-up.
* having at least 3 symptoms of hypoglycemia presented in the dumping severity scale (DSS).
* at least one of these symptoms must be a neuroglycopenic symptom
* all these symptoms have an intensity of 2 or 3 on DSS.

Exclusion Criteria:

* severe surgery-related complication
* revisional surgery
* life threatening health conditions.
* diabetes mellitus or other metabolic diseases
* pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
blood sugar variation | 4 weeks
  measured by continuous blood glucose monitor

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Landstad, phd, Study Director — Helse Nord-Trøndelag HF
Locations (1):
- Obesity Outpatient Clinic, Surgical Clinic, Nord-Trøndelag Hospital Trust, Hospital of Namsos, Namsos, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: No